CLINICAL TRIAL: NCT04174339
Title: PD-1 Antibody(SHR-1210) Plus Apatinib Combined With POF in Treatment Naive Advanced Gastric Cancer: A Phase II Study.
Brief Title: PD-1 Antibody(SHR-1210) Plus Apatinib Combined With POF in Advanced Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNF-017
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-10

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — camrelizumab; spartalizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab plus apatinib and POF (Experimental): Participants will receive camrelizumab in combination with apatinib plus POF until pre-defined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate; Drug: POF

INTERVENTIONS:
Drug: Camrelizumab — Subjects receive SHR-1210 intravenously, Dosage form: lyophilised powder, Strength: 200 mg /vial，d1
  Other Names: SHR-1210; PD-1 Antibody
Drug: Apatinib Mesylate — Subjects receive Apatinib orally, Dosage form: tablet, Strength: 250 mg/tablet，TID
Drug: POF — The POF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.

SUMMARY:
This study is a single center, phase II study, to evaluate the effectiveness and safety of PD-1 Antibody(SHR-1210) Plus apatinib Combined With POF(paclitaxel plus oxaliplatin plus 5-fluorouracil plus leucovorin) , in the first-line treatment for patients with advanced/metastatic gastric cancer.

DETAILED DESCRIPTION:
This is a exploratory, single-arm, open-label trial. The investigator's primary purpose is to compare that ORR of patients with camrelizumab plus apatinib and POF for advanced/metastatic gastric cancer.

In treatment period, patients will be administrated camrelizumab plus apatinib and POF, every 28 days for 1 cycle, until disease progression, toxicity intolerance, withdrawal of informed consent, patients judged must be terminated study termination.

The imaging evaluation was performed according to the RECIST 1.1 criteria every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced unresectable, histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.
2. No previous treatment with chemotherapy or radiation therapy.
3. Ability to take medications orally.
4. With measurable lesions,according to Response Evaluation Criteria In Solid Tumors Version 1.1.
5. Patients must have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
6. Without serious system dysfunction and could tolerate chemotherapy. With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a leucopenia count of ≥4.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.
7. Life expectancy ≥3 months.
8. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
9. With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

1. Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
2. With any acitve autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatititis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
3. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents: systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
4. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), orventricular arrhythmia which need medical intervention.
5. Known history of hypersensitivity to any components of the SHR-1210 formulation, or other antibody formulation.
6. Prior systemic chemotherapy, radiotherapy, immunotherapy, hormone therapy, surgery or target therapy within 4 weeks.
7. Coagulation abnormalities (PT>16s、APTT>43s、TT>21s、Fbg<2g/L), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
8. Has known active central nervous system metastatases.
9. Pregnant (positive pregnancy test) or breast feeding.
10. History of a stroke or CVA within 6 months. Clinically significant peripheral vascular disease.
11. Inability to comply with study and/or follow-up procedures. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-10 (Estimated); Primary Completion 2020-12-09 (Estimated); Study Completion 2021-05-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From enrollment to 12 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | From enrollment to 12 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
  The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.
Overall Survival (OS) | From enrollment to 12 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
  The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Disease control rate(DCR) | From enrollment to 12 month
  DCR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR or SD. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR or SD to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Rongbo Lin, Fuzhou, China